CLINICAL TRIAL: NCT02854852
Title: Accuracy of Photoplethysmography to Detect Changes in Vascular Tone: a Doppler Study
Brief Title: Photoplethysmography Detects Changes in Vascular Tone
Status: Completed | Type: Observational
Sponsor: Hospital Privado de Comunidad de Mar del Plata (Other)
Responsible Party: Sponsor
Other Study IDs: 359/16
Record Dates: First submitted 2016-08-01; First posted 2016-08-04 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-01

CONDITIONS: Vascular Diseases
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients undergoing general anesthesia: Patients ASA 1-3, undergoing different types of general anesthesia, in supine position, with standard or advanced hemodynamic monitoring.

SUMMARY:
Changes in the vascular tone of anesthetized patients is common and cause hemodynamic problems. The monitoring of such changes in vascular resistance using simple and non-invasive tools is lacking. The present study was designed to determine if photoplethysmography can detect changes in the systemic vascular resistance using Doppler as the reference method.

DETAILED DESCRIPTION:
This is a prospective and observational study designed to test the reliability of photoplethysmography to diagnose changes in the vascular resistance during anesthesia. The investigators will studied 50 mechanically ventilated patients undergoing general anesthesia. Photoplethysmography will be continuously recorded in the right thumb during anesthesia. Duplex color and power Doppler will measure flow in the radial artery of the right hand.The contour analysis of both, photoplethysmogram and radial artery flow will be analyzed, correlated and compared using the Bland-Altman plot.

ELIGIBILITY:
Inclusion Criteria:

* Written Inform Consent
* Programmed surgery
* Supine position

Exclusion Criteria:

* Emergency surgery
* Peripheral vascular diseases

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2018-01-22 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Accuracy of photoplethysmography for the assessment of systemic vascular tone | 5 hours
  Comparison between pletysmography with the reference Doppler method

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Tusman, MD, Principal Investigator — Study Principal Investigato
Locations (1):
- Hospital Privado de Comunidad, Mar del Plata, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No